CLINICAL TRIAL: NCT06085339
Title: Social Media Use in Adolescent Diabetes Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004205
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Media Exposure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Media Intervention (Experimental): In addition to receiving usual care, participants enrolled in the social media arm will receive diabetes education and support over the course of 6 months by following the study team's Instagram page and engaging with the study team and other adolescent participants on Instagram.
  Interventions: Behavioral: Social Media
- Usual Care (No Intervention): Usual care reflects the standard treatment currently provided to adolescents living with type 1 diabetes. Every adolescent with diabetes is cared for by a team of diabetes specialists which includes a provider (MD, Physician Assistant and/or Nurse Practitioner), registered nurse, nutritionist and social worker. Adolescents with type 1 diabetes are seen by their multidisciplinary team approximately every 3 months. In addition, they have access to their multidisciplinary care team via telephone and/or MyChart communication as often as is necessary between clinic visits.

INTERVENTIONS:
Behavioral: Social Media — The social media arm participants will receive a diabetes curriculum designed to address diabetes self-efficacy and independence with diabetes management over the course of 6 months. Participants will have the option to engage with the study team and other participants through Instagram posts and direct messaging.
  Arms: Social Media Intervention

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of a social media intervention to support diabetes management in adolescents with type 1 diabetes.

Adolescent participants will be randomized to receive diabetes education and peer support over Instagram or to usual outpatient diabetes care. Researchers will assess whether the social media intervention is feasible. In addition, the study team will also explore and compare changes in glucose levels and person-reported outcomes between the two groups.

DETAILED DESCRIPTION:
The majority of adolescents with type 1 diabetes do not meet recommended glycemic targets, placing them at risk for acute and chronic diabetes-related complications. Strategies that improve adolescent diabetes self-management are needed. Social media offers new opportunities to provide diabetes education and peer support through communication in a digital environment.

As part of a randomized controlled trial, adolescent participants will be randomized to receive diabetes education and peer support over Instagram in addition to usual care or to standard outpatient diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes ≥12 months
* Most recent hemoglobin A1c (HbA1c) level is > 7.0%
* Currently use Dexcom continuous glucose monitoring (CGM) system
* Speak English fluently
* Cognitively able to participate in program on Instagram and complete surveys
* Have access to a personal Instagram account
* Found to be eligible on the Social Media Preference Screener

Exclusion Criteria:

* Patient is a ward of the state
* Patient is pregnant as diabetes standard of care is different during pregnancy (i.e., different glycemic targets and frequency of clinic visits)
* Severe comorbidities including other major chronic health conditions that significantly impact daily management demands or health outcomes

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Enrollment | 0 months
  Percentage of participants who enroll in study after in-person or remote discussion about study participation.
Feasibility: Retention Rate | 6 months
  Percentage of enrolled participants who complete the final 6-month surveys.

SECONDARY OUTCOMES:
Hemoglobin A1c (HbA1c) | Change over 6 months
  HbA1c laboratory measurements collected during the intervention.
Time In Range | Change over 6 months
  Continuous glucose monitor sensor glucose measurements collected during the intervention that are in range (70-180 mg/dL).
Time Above Range | Change over 6 months
  Continuous glucose monitor sensor glucose measurements collected during the intervention that are above range (>180 mg/dL).
Time Below Range | Change over 6 months
  Continuous glucose monitor sensor glucose measurements collected during the intervention that are below range (<70 mg/dL).
Diabetes Self-Management | Change over 6 months
  Adherence will be assessed with the Diabetes Self-Management Questionnaire. Higher scores indicate higher adherence to diabetes self-management.
Diabetes Distress | Change over 6 months
  Diabetes distress will be assessed with the Problem Areas in Diabetes Scale -- Teen Version. Higher scores indicate higher diabetes distress.
Diabetes Family Conflict | Change over 6 months
  Diabetes family conflict will be assessed with the Diabetes Family Conflict Scale. Higher scores indicate higher diabetes family conflict.
Health Care Transition Readiness | Change over 6 months
  Health care transition readiness will be assessed with the Readiness Assessment in Emerging Adults with Type 1 Diabetes Diagnosed in Youth. Higher scores indicate higher health care transition readiness.
Depressive Symptoms | Change over 6 months
  Depressive symptoms will be assessed with the Patient Health Questionnaire-8. Higher scores indicate higher depressive symptoms.
Mental Wellbeing | Change over 6 months
  Mental wellbeing will be assessed with the Warwick-Edinburgh Mental Wellbeing Scale. Higher scores indicate higher mental wellbeing.
Problematic Internet Use | Change over 6 months
  Adolescent problematic internet use will be assessed with the Problematic and Risky Internet Use Screening Scale. Higher scores indicate higher concern for problematic internet use.
Diabetes Strengths | Change over 6 months
  Adolescents' diabetes-specific "strengths" (i.e., positive behaviors and attitudes related to the challenges of living with type 1 diabetes) will be assessed with the Diabetes Strengths and Resilience measure. Higher scores indicate increased diabetes-specific strengths.
Diabetes Quality of Life | Change over 6 months
  Diabetes-specific quality of life will be assessed using the adolescent self-report version of the Type 1 Diabetes and Life. Higher scores indicate higher diabetes-specific quality of life.
Screen Time | Change over 6 months
  Screen time use will be measured by the Screen Time summary from a participant's smartphone device.

CONTACTS AND LOCATIONS:
Overall Officials: Faisal S Malik, MD, MSHS, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided